CLINICAL TRIAL: NCT02866188
Title: The Feasibility Study of Recognition of Cardiac Arrest Using a Smart Watch
Acronym: TFSRCASW
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hanyang University (Other)
Responsible Party: Principal Investigator, LEE YOON-JE, Emergency physician, Hanyang University
Other Study IDs: SWROCA
Record Dates: First submitted 2016-08-10; First posted 2016-08-15 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-08

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Check pulse with Smart watch on 3 parts of patient's body surface — Check pulse with smart watch on wrist, carotid artery, and eye of patients in shock or cardiac arrest state.

SUMMARY:
In this study, we want to find out whether the recognition of cardiac arrest using a smart watch is feasible or not. If this idea is possible, the recognition of cardiac arrest using the smart watch is easy and fast to the witness, like a general person. By using the smart watch, the emergency response system for cardiac arrest and the bystander CPR or BLS is beginning earlier than using conventional cardiac arrest recognition method in field.

DETAILED DESCRIPTION:
In Korea, an out-of-hospital cardiac arrest (OHCA) was occurred twenty thousand person per year, and among them sixty percent was occurred in their home. We already knew that a survivor rate and neurological outcome of OHCA patient has a close relation with initial emergency management in field, like a bystander cardiopulmonary resuscitation (CPR), Basic Life Support (BLS), etc. However, in Korea, a witness almost did not the bystander CPR or BLS in field until highly trained rescuers arrived there. So, total survivor rate is just 2.4 % irrespective of neurologic outcome in Korea.

Generally, in Korea, a beginning of the bystander CPR progress throughout dispatcher's instruction of emergency response system. This system for OHCA patient activate only when the witness recognize cardiac arrest and call the emergency response system. Therefore, cardiac arrest recognition by the witness is very important.

However, a conventional recognition of cardiac arrest in field is often difficult, because there are no monitoring devices, healthcare providers. The conventional recognition method of cardiac arrest is that it is firstly to check mental status, secondly check pulse on patient's carotid artery and self-respiration. This method is too difficult for the witness, especially general persons. Even, it is difficult for an emergency physicians, too.

Consequentially, the recognition of cardiac arrest by the witness is generally delayed, a golden-time is running out until highly trained rescuers arrive there. An average arrival time of highly trained rescuers is eight to ten minutes. A hypoxic brain damage is begin from four minutes after cardiac arrest. As a result, this delayed time is already passed four minutes after cardiac arrest. So, the survivor rate and the neurologic outcome are not good enough.

In this study, we want to find out whether the recognition of cardiac arrest using a smart watch is feasible or not. If this idea is possible, the recognition of cardiac arrest using the smart watch is easy and fast to the witness, like a general person. By using the smart watch, the emergency response system for cardiac arrest and the bystander CPR or BLS is beginning earlier than using conventional cardiac arrest recognition method in field.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Shock
* Cardiac arrest

Exclusion Criteria:

* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Shock or Cardiac arrest patients in emergency room.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-08; Primary Completion 2016-11 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
The minimum blood pressure on wrist | 10 seconds
  mmHg, Blood pressure in minimum checkable pulse using smart watch
The minimum blood pressure on carotid artery | 10 seconds
  mmHg, Blood pressure in minimum checkable pulse using smart watch
The minimum blood pressure on eye | 10 seconds
  mmHg, Blood pressure in minimum checkable pulse using smart watch

CONTACTS AND LOCATIONS:
Locations (1):
- Hanyang University Guri Hospital, Guri-si, Gyeonggi-do, South Korea